CLINICAL TRIAL: NCT03489486
Title: MET: REevaluation for Perioperative cArdIac Risk (MET-REPAIR): a Prospective, Multi-centre Cohort Observational Study- Presepsin (sCD14-ST) for Perioperative Risk Prediction Nested Cohort Study
Brief Title: Presepsin (sCD14-ST) for Prediction of Perioperative Risk - MET-REPAIR Nested Cohort Study
Acronym: P^3-MET-REPAIR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Collaborators: European Society of Anaesthesiology (Other)
Responsible Party: Principal Investigator, Jan Larmann, Dr., PhD, University Hospital Heidelberg
Other Study IDs: MET-REPAIR PRESEPSIN
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Non Cardiac Surgery
Keywords: Presepsin; sCD14-ST; biomarker; perioperative risk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicentre international prospective cohort study designed to evaluate whether preoperative presepsin (sCD14-ST) is associated with the composite endpoint: all-cause mortality and major adverse cardiovascular or cerebrovascular events (MACCE) after elevated risk non-cardiac surgery. If so:

1. What is the optimal cut-off for presepsin to predict the composite endpoint all-cause mortality and MACCE?
2. Does the calculated optimal cut-off improve prediction of the composite endpoint all-cause mortality and MACCE when added to clinical data and established biomarkers?

DETAILED DESCRIPTION:
Major non-cardiac surgery is still associated with relevant cardiovascular mortality and morbidity. In Europe, in-hospital mortality exceeded 7% in patients with coronary artery disease and in those with congestive heart failure. Within 30 days of non-cardiac surgery procedures, 8% of patients will suffer a major cardiovascular event.

Immunological processes, increased recruitment and infiltration of innate and adaptive immune cells into atherosclerotic lesions, have been shown to drive perioperative atherosclerotic lesion progression and plaque destabilization and are thought to promote plaque rupture. When classical monocytes are activated to inflammatory non-classical monocytes, the membrane-bound cell surface protein CD14 is released into circulation. In plasma, soluble CD14 (sCD14) is cleaved by lysosomal proteases. The N-terminal 13kDa fragment constitutes sCD14 subtype (sCD14-ST), also called presepsin. Presepsin has been established as a marker for early identification of patients with systemic infections. Recently, presepsin has been proposed as a biomarker for preoperative risk prediction in cardiac surgery. Our preliminary results in a limited number of patients suggest that presepsin is associated with major adverse cardiovascular and cerebrovascular events after non-cardiac surgery as well with all-cause mortality. Presepsin might have a test characteristic superior to conventional risk assessment on the basis of the revised cardiac risk index (RCRI), high-sensitivity cardiac Troponin-T (hs-cTnT) and N-terminal prohormone of brain natriuretic peptide (NT-proBNP).

Preoperative presepsin quantification might help to identify non-cardiac surgery patients prone to experience perioperative major adverse cardiovascular and cerebrovascular events.

ELIGIBILITY:
Inclusion criteria:

* Enrollment in MET-REPAIR (NCT03016936)
* Signed written informed consent

No exclusion criteria

I

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective, elevated-risk noncardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1695 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Composite of intra- and postoperative in hospital all-cause mortality, non-fatal cardiac arrest, acute myocardial infarction, congestive heart failure requiring transfer to a higher unit of care or prolonging stay on ICU/intermediate care ≥24h and stroke | at discharge or at day 30 after surgery (whatever comes first)
  Number of Patients with Composite of intra- and postoperative in hospital all-cause mortality, non-fatal cardiac arrest, acute myocardial infarction, congestive heart failure requiring transfer to a higher unit of care or prolonging stay on ICU/intermediate care ≥24h and stroke

SECONDARY OUTCOMES:
Composite of intra- and postoperative in hospital all-cause mortality, non-fatal cardiac arrest, acute myocardial infarction, congestive heart failure requiring transfer to a higher unit of care or prolonging stay on ICU/intermediate care ≥24h and stroke | 30 days
  Number of Patients with composite of intra- and postoperative in hospital all-cause mortality, non-fatal cardiac arrest, acute myocardial infarction, congestive heart failure requiring transfer to a higher unit of care or prolonging stay on ICU/intermediate care ≥24h and stroke for patients recruited in centers conducting 30-day follow-up
All-cause mortality | 30 days
  Number of patients that die of any cause
Non-fatal cardiac arrest | 30 days
  Number of patients with non-fatal cardiac arrest
Myocardial infarction | 30 days
  Number of patients with myocardial infarction
Congestive heart failure requiring transfer to a higher unit of care or prolonging stay on ICU/intermediate care (≥24h) | 30 days
  Number of patients with congestive heart failure requiring transfer to a higher unit of care or prolonging stay on ICU/intermediate care (≥24h)
Stroke | 30 days
  Number of patients with stroke
Cardiovascular mortality | 30 days
  Number of patients that die of a cardiovascular cause
In-hospital cardiovascular mortality | 30 days
  Number of patients that die in hospital of a cardiovascular cause
Complications ≥ 3 in Clavien Dindo Classification | within 30 days after surgery
  Number of patients with ≥ 3 complications in Clavien Dindo Classification
Length of Hospital stay | within 30 days after surgery
  Number of days participants stayed in hospital
Length of ICU stay | within 30 days after surgery
  Number of days participants stayed in ICU
Myocardial injury after non-cardiac surgery (MINS) | within 30 days after surgery
  Number of Patients with MINS

CONTACTS AND LOCATIONS:
Overall Officials: Jan Larmann, MD/PhD, Principal Investigator — Department of Anesthesiology, Univeristy Hospital Heidelberg
Locations (1):
- Department of Anaesthesiology, University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Background] Devereaux PJ, Mrkobrada M, Sessler DI, Leslie K, Alonso-Coello P, Kurz A, Villar JC, Sigamani A, Biccard BM, Meyhoff CS, Parlow JL, Guyatt G, Robinson A, Garg AX, Rodseth RN, Botto F, Lurati Buse G, Xavier D, Chan MT, Tiboni M, Cook D, Kumar PA, Forget P, Malaga G, Fleischmann E, Amir M, Eikelboom J, Mizera R, Torres D, Wang CY, VanHelder T, Paniagua P, Berwanger O, Srinathan S, Graham M, Pasin L, Le Manach Y, Gao P, Pogue J, Whitlock R, Lamy A, Kearon C, Baigent C, Chow C, Pettit S, Chrolavicius S, Yusuf S; POISE-2 Investigators. Aspirin in patients undergoing noncardiac surgery. N Engl J Med. 2014 Apr 17;370(16):1494-503. doi: 10.1056/NEJMoa1401105. Epub 2014 Mar 31. PMID 24679062
- [Background] Kristensen SD, Knuuti J, Saraste A, Anker S, Botker HE, De Hert S, Ford I, Gonzalez Juanatey JR, Gorenek B, Heyndrickx GR, Hoeft A, Huber K, Iung B, Kjeldsen KP, Longrois D, Luescher TF, Pierard L, Pocock S, Price S, Roffi M, Sirnes PA, Uva MS, Voudris V, Funck-Brentano C; Authors/Task Force Members. 2014 ESC/ESA Guidelines on non-cardiac surgery: cardiovascular assessment and management: The Joint Task Force on non-cardiac surgery: cardiovascular assessment and management of the European Society of Cardiology (ESC) and the European Society of Anaesthesiology (ESA). Eur J Anaesthesiol. 2014 Oct;31(10):517-73. doi: 10.1097/EJA.0000000000000150. No abstract available. PMID 25127426
- [Background] Fleisher LA, Fleischmann KE, Auerbach AD, Barnason SA, Beckman JA, Bozkurt B, Davila-Roman VG, Gerhard-Herman MD, Holly TA, Kane GC, Marine JE, Nelson MT, Spencer CC, Thompson A, Ting HH, Uretsky BF, Wijeysundera DN; American College of Cardiology; American Heart Association. 2014 ACC/AHA guideline on perioperative cardiovascular evaluation and management of patients undergoing noncardiac surgery: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines. J Am Coll Cardiol. 2014 Dec 9;64(22):e77-137. doi: 10.1016/j.jacc.2014.07.944. Epub 2014 Aug 1. No abstract available. PMID 25091544
- [Background] Lee TH, Marcantonio ER, Mangione CM, Thomas EJ, Polanczyk CA, Cook EF, Sugarbaker DJ, Donaldson MC, Poss R, Ho KK, Ludwig LE, Pedan A, Goldman L. Derivation and prospective validation of a simple index for prediction of cardiac risk of major noncardiac surgery. Circulation. 1999 Sep 7;100(10):1043-9. doi: 10.1161/01.cir.100.10.1043. PMID 10477528
- [Background] Gupta PK, Gupta H, Sundaram A, Kaushik M, Fang X, Miller WJ, Esterbrooks DJ, Hunter CB, Pipinos II, Johanning JM, Lynch TG, Forse RA, Mohiuddin SM, Mooss AN. Development and validation of a risk calculator for prediction of cardiac risk after surgery. Circulation. 2011 Jul 26;124(4):381-7. doi: 10.1161/CIRCULATIONAHA.110.015701. Epub 2011 Jul 5. PMID 21730309